CLINICAL TRIAL: NCT05831293
Title: The Effect of Mindfulness Based Stress Reduction Program on Stress and Quality of Life in Family Caregivers of Patients With Cancer: Randomized Controlled Trial
Brief Title: Mindfulness-Based Reduction Stress Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, NİHAN TÜRKOĞLU, Assist Prof., Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: nihann
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-11

CONDITIONS: Cancer; Caregiver Stress; Quality of Life
MeSH Terms: conditions — Neoplasms; Caregiver Burden

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): In each session, three sections were discussed and reviewed: (1) last week's experiences, (2) training, and (3) practice. Each session usually began with mindfulness and meditation exercises, followed by group discussion, review of homework activities, and introduction to new exercises. Participants were asked to complete 15-30 minutes of daily practice each week.
  Interventions: Behavioral: Mindfulness Based Stress Reduction Program
- Control (No Intervention): No intervention will be applied to the control group.

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction Program — In each session, three sections were discussed and reviewed: (1) last week's experiences, (2) training, and (3) practice. Each session usually began with mindfulness and meditation exercises, followed by group discussion, review of homework activities, and introduction to new exercises. Participants were asked to complete 15-30 minutes of daily practice each week.
  Arms: Experimental

SUMMARY:
The participants consisted of 1332 caregivers of patients diagnosed with cancer, who applied to Atatürk University Health Research and Application Center, Outpatient Chemotherapy Unit between December 2022 and March 2023. In the power analysis, the sample of the research; According to Cohen, a total of 108 people, 54 of whom were in the experimental group and 54 in the control group, with a medium effect size of 0.5%, an error margin of 0.05% and a confidence interval of 0.95%, were 95% representative of the universe. Against the possibility of data loss, 20% backup sample was included in this number and the study was planned with a total of 124 people, 62 in the experimental group and 62 in the control group. 20 participants were excluded on the basis of inclusion and exclusion criteria. 104 participants formed the sample

DETAILED DESCRIPTION:
Pretest measurements (T1) were made to the individuals in the experimental and control groups. 8-week mindfulness-based interventions were administered online to caregivers of cancer patients (Table 1). Before starting the MDI program in the experimental group, visual and written materials about the sessions prepared by the researchers were distributed. The program was implemented 4 days a week, 1 session a day, and each session was implemented in groups of 10-15 people for 60-90 minutes. After the 8-week MDI Program of the experimental group was completed, the data collection forms were re-applied to the individuals in the experimental and control groups, and posttest-1 measurements (T2) were made. 4 weeks after the posttest-1 measurements, the posttest-2 measurements (T3) of the individuals in the experimental and control groups were performed.

ELIGIBILITY:
Inclusion Criteria:

* No psychiatric problems,
* Over 18,
* literate,
* Having internet access at home,
* Not receiving or planning to receive therapy support during the education process,
* Not having any previous mindfulness experience

Exclusion Criteria:

* Those who want to leave the study,
* Do not accept to participate in the research
* not at a level to answer the questions asked cognitively.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Caregiver Stress Scale | two week
  The scale was developed by Robinson (1983) to measure the subjective care burden of caregivers and to quickly identify families with care concerns. Its Turkish adaptation was made by Uğur and Fadıloğlu (2006). The reliability coefficient of the scale was found to be 0.77. The scale consists of 13 items. The scoring of the scale is between 0-1. A score above 7 indicates the burden of care subjectively.
The Caregiver Quality of Life Index Cancer Scale -CQOLC | Two week
  It was developed by Weitzner et al. to measure the quality of life of caregivers of cancer patients, including physical function, emotional function, family function, and social function. The total score of each sub-dimension and scale in the scale varies between 0 and 140. A higher score indicates a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Nihan Türkoğlu, Assist.Prof., Study Chair — Ataturk University
Locations (1):
- Ataturk Unıversity, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No